CLINICAL TRIAL: NCT00150943
Title: The Benefit of STent Placement and Blood Pressure and Lipid-Lowering for the Prevention of Progression of Renal Dysfunction Caused by Atherosclerotic Ostial Stenosis of the Renal Artery (STAR)
Brief Title: Stenting in Renal Dysfunction Caused by Atherosclerotic Renal Artery Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C99.1810-STAR; C99.1810
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Renal Artery Obstruction; Kidney Failure
Keywords: Renal artery stenosis; Stent; Renal failure; Atorvastatin; Hypertension; Atherosclerosis
MeSH Terms: conditions — Renal Artery Obstruction; Renal Insufficiency; Hypertension; Atherosclerosis

INTERVENTIONS:
Device: Renal artery stent

SUMMARY:
Background:

Atherosclerotic renal artery stenosis (ARAS) is associated with progressive loss of renal function and is one of the most important causes of renal failure in the elderly. Current treatment includes restoration of the renal arterial lumen by endovascular stent placement. However, this treatment only affects damage caused by ARAS due to the stenosis and ensuing post-stenotic ischemia. ARAS patients have severe general vascular disease. Atherosclerosis and hypertension can also damage the kidney parenchyma causing renal failure. Medical treatment focuses on the latter. Lipidlowering drugs (statins) could reduce renal failure progression and could reduce the overall high cardiovascular risk. The additional effect on preserving renal function of stent placement as compared to medical therapy alone is unknown. Therefore, the STAR-study aims to compare the effects of renal artery stent placement together with medication vs. medication alone on renal function in ARAS patients.

Method:

Patients with an ARAS of ≥50% and renal failure (creatinine (Cr) clearance <80 mL/min/1.73 m2) are randomly assigned to stent placement with medication or to medication alone. Medication consists of statins, anti-hypertensive drugs and antiplatelet therapy. Patients are followed for 2 yrs with extended follow-up to 5 yrs. The primary outcome of this study is a reduction in Cr clearance >20% compared to baseline. This trial will include 140 patients.

DETAILED DESCRIPTION:
This is a randomized, multicenter trial of patients with an ostial ARAS and renal failure. Patients will be randomized to:

(i)medical treatment consisting of antihypertensive, lipid-lowering and antiplatelet therapy plus the advice to stop smoking; or (ii)medical treatment as outlined in (i) with additional stent placement.

Patients with an ostial ARAS, a Cr clearance of <80 mL/min/1.73m2 according to the Cockcroft and Gault formula and stable blood pressure (BP) control are enrolled in this trial. Ostial ARAS is defined as a luminal reduction of ≥50% of the renal artery within 1 cm of the aortic wall, in the presence of atherosclerotic changes of the aorta. Stenosis evaluation can be performed on CT-angiography, MR angiography or intra-arterial angiography.

Medical therapy: Irrespective of baseline serum cholesterol values, the patients will be treated with lipid-lowering therapy: 10 mg of atorvastatin and if this is well tolerated the dose will be doubled to the final dose of 20 mg. Any lipid-lowering medication currently used is discontinued and replaced by atorvastatin. Hypertension is treated with the following drugs: thiazide diuretic, calcium antagonist, beta-blocker and alpha-blocker. ACE-inhibitors/angiotensin-II-antagonists together with increasing loop diuretic doses, should be used only as a last resort antihypertensive treatment when other classes of antihypertensive agents have failed. The target BP is <140/90 mmHg. Patients will receive anti-platelet therapy, aspirin 75-100 mg/od. Considering that smoking is a major renal risk factor, smokers will be advised to stop.

Stent and medical therapy: Medical therapy is identical in the two treatment arms. In the stent group, patients will start with aspirin 75-100 mg/od the day before admission. The stent (Palmaz-Corinthian IQ/Palmaz Genesis, Johnson & Johnson Medical, NV/SA) will be placed during an in-patient admission according to a standardized protocol.

Randomisation will be done per participating centre and will be stratified for unilateral or bilateral abnormalities. An unilateral abnormality is defined as an unilateral ostial stenosis and on the other side a normal renal artery or a truncal stenosis (a truncal stenosis is nearly always easy to dilate by angioplasty). All other patients are considered to have bilateral abnormalities

Clinical follow-up is scheduled after 1, 3 and then every 3 months for the first 2 yrs and every 6 months until the 5 yr follow-up is completed. Economic data are assessed after 3 mths and every 3 mths for 2 yrs. Quality of life will be measured by standardized SF-36 and EQ-5D health questionnaires before, after 1 mth and every 6 mths for 2 yrs.

Indications for stent placement in the medically treated patients and re-angiography and balloon dilatation of the stent in the stented patients are: (i) a persistent >20% reduction of Cr clearance; (ii) therapy refractory hypertension (defined as an office BP >180/100 mmHg during three follow-up visits and subsequently a mean daily BP of >160/95 mmHg on 24 hr ambulant BP monitoring, while on the maximum dose of all classes of antihypertensives); (iii) pulmonary edema in the presence of bilateral renovascular disease and a normal or slightly impaired left ventricular function on echocardiography in combination with ACE-inhibitors/angiotensin-II antagonist intolerance defined as a fall of estimated Cr clearance by >20% and; (iv) malignant hypertension (defined as fundus grade III/IV).

Analysis of results: The difference in the proportion of patients with progressive renal dysfunction between both treatment arms will be assessed including 95% confidence intervals (95% CI). Mean change and difference in renal function change, including 95% CI will be reported. With multivariate logistic regression analysis not only will the effects of the two treatment strategies be evaluated, but also whether there are independent effects of age, smoking, proteinuria, bilateral or unilateral renal artery stenosis, BP and renal function at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ostial atherosclerotic renal artery stenosis ≥50% on CTA, MRA or intra-arterial angiography
* Estimated creatinine clearance <80 ml/min/1.73m2 according to the Cockcroft and Gault formula, on two occasions within one month

Exclusion Criteria:

* Declined informed consent
* Proven cholesterol embolisation at previous interventions
* Renal artery diameter <4mm
* Estimated creatinine-clearance <15ml/min/1.73m2
* Diabetes Mellitus with proteinuria >3g/24h
* Any known cause of renal failure other than ischemic nephropathy
* Pulmonary oedema in the presence of bilateral renovascular disease in combination with intolerance of ACE-inhibitors/ Angiotensin-II antagonists defined as a fall of estimated creatinine clearance of >20%
* Malignant hypertension (fundus grade III/IV)
* Myocardial infarction or CVA <3 months before planned date of inclusion
* Contra-indication for the use of atorvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2000-06

PRIMARY OUTCOMES:
Progressive renal function loss (= reduction in estimated Cr clearance by >20%) after 2 yrs follow-up, with an extended follow-up of 5 yrs

SECONDARY OUTCOMES:
Acute complications
Late complications
Occlusion of the stenotic renal artery
Incidence and time to doubling of serum Cr
Initiation of dialysis therapy
Effect on hypertension and the occurrence of therapy refractory or malignant hypertension
Incidence of pulmonary edema
Cardiovascular morbidity and mortality
Total mortality
Cost-effectiveness
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jaap J. Beutler, MD.PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Bax L, Mali WP, Buskens E, Koomans HA, Beutler JJ, Braam B, Beek FJ, Rabelink TJ, Postma CT, Huysmans FT, Deinum J, Thien T, Schultze Kool LJ, Woittiez AJ, Kouwenberg JJ, van den Meiracker AH, Pattynama PM, van de Ven PJ, Vroegindeweij D, Doorenbos CJ, Aarts JC, Kroon AA, de Leeuw PW, de Haan MW, van Engelshoven JM, Rutten MJ, van Montfrans GA, Reekers JA, Plouin PF, La Batide Alanore A, Azizi M, Raynaud A, Harden PN, Cowling M; STAR Study Group. The benefit of STent placement and blood pressure and lipid-lowering for the prevention of progression of renal dysfunction caused by Atherosclerotic ostial stenosis of the Renal artery. The STAR-study: rationale and study design. J Nephrol. 2003 Nov-Dec;16(6):807-12. PMID 14736007
- [Derived] Bax L, Woittiez AJ, Kouwenberg HJ, Mali WP, Buskens E, Beek FJ, Braam B, Huysmans FT, Schultze Kool LJ, Rutten MJ, Doorenbos CJ, Aarts JC, Rabelink TJ, Plouin PF, Raynaud A, van Montfrans GA, Reekers JA, van den Meiracker AH, Pattynama PM, van de Ven PJ, Vroegindeweij D, Kroon AA, de Haan MW, Postma CT, Beutler JJ. Stent placement in patients with atherosclerotic renal artery stenosis and impaired renal function: a randomized trial. Ann Intern Med. 2009 Jun 16;150(12):840-8, W150-1. doi: 10.7326/0003-4819-150-12-200906160-00119. Epub 2009 May 4. PMID 19414832